CLINICAL TRIAL: NCT02271256
Title: Safety and Efficacy of Functional Intimate Apparel for Adolescents With Early Scoliosis
Brief Title: Functional Intimate Apparel for Adolescents With Early Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Joanne Yip, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRF2015
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Scoliosis
Keywords: Functional intimate apparel; Adolescent Idiopathic scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Intervention Model Description: There are 2 groups of subjects. One group receives the treatment of functional intimate apparel which is called FIA group while one group receives observation only, which is called control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional intimate apparel (Experimental): A functional intimate apparel will be provided to patient to wear it 8 hours daily. Monitoring and observation will be provided during the 6-9 months wearing period.
  Interventions: Device: Functional Intimate Apparel
- Control (No Intervention): Monitoring and observation will be provided during the 6-9 months wearing period.

INTERVENTIONS:
Device: Functional Intimate Apparel — The design of functional intimate apparel will incorporate different mechanisms, such as a) compression and pulling forces through a close fit of the intimate apparel, b) lumbar flexion by using a supporting belt, c) transverse forces applied by inserting pads inside the pocket lining with the application of 3-point pressure system, d) axial rotation or coupled motion by using uneven straps, and e) an active mechanism that aims to shift the trunk away from areas of pressure.
  Arms: Functional intimate apparel

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a prevalent chronic condition that gradually leads to the three dimensional deformity of the spine. Spinal curvature increases in youths as puberty progresses. Generally, only observation is suggested for adolescents with early scoliosis (Cobb's angle ≤ 20°). Rigid brace treatment is too draconian for them due to the high corrective force which nearly constrains all movements. Flexible brace treatment is an alternative; however, its efficacy is still controversial. Functional intimate apparel with a specialized design for teenagers with scoliosis is limited and most part of them can only provide some improvement for bad postures, such as hunchback. A scientific approach should be used to design and develop functional intimate apparel as a treatment option for adolescents with early scoliosis.

This project aims to combine clinical experience with textiles and materials sciences to research and develop a functional intimate apparel for adolescents with early scoliosis. As a result, this will reduce the future likelihood of brace wear or surgery.

In this study, the eligible subjects will be given a functional intimate apparel to wear for 8 hours a day. Monitoring and observation will be provided during a 6-month wear trial. The effectiveness of the functional intimate apparel will be evaluated by pre- and post- treatment X-ray radiography and sonography.

DETAILED DESCRIPTION:
This project aims to combine clinical experience with textiles and materials sciences to research and develop a functional intimate apparel for adolescents with early scoliosis. As a result, this will reduce the future likelihood of brace wear or surgery.

The design of functional intimate apparel will incorporate different mechanisms, such as a) compression and pulling forces through a close fit of the intimate apparel, b) lumbar flexion by using a supporting belt, c) transverse forces applied by inserting pads inside the pocket lining with the principle of the 3-point pressure system, d) axial rotation or coupled motion by using a system with uneven straps, and e) an active mechanism that aims to shift the trunk away from areas of pressure.

In this study, the eligible subjects will be given a functional intimate apparel to wear for 8 hours a day. Monitoring and observation will be provided during a 6-month wear trial. The effectiveness of the functional intimate apparel will be evaluated by pre- and post- treatment X-ray radiography and sonography.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 to 13 years
* Diagnosis of AIS in early stage
* Primary Cobb angle 15-35 degrees
* Pre-menarche or post- menarche by no more than 1 year
* Ability to read and understand English or Chinese
* At high risk for curve progression
* Skeletally immature (Risser grade 0,1 or 2)
* Physical and mental ability to adhere to functional intimate apparel protocol

Exclusion Criteria:

* Contraindications for x-ray exposure
* Diagnosis of other musculoskeletal or developmental illness that might be responsible for the spinal curvature
* History of previous surgical or orthotic treatment for AIS
* Contraindications for pulmonary and/ or exercise tests
* Psychiatric disorders
* Recent trauma
* Recent traumatic (emotional) event

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Instant spinal correction | 2 hours after wearing the functional intimate apparel
  Measure lateral curvature of vertebra under x-ray. The instant effectiveness of the functional intimate apparel will be evaluated through radiography.
Six-month spinal control | 6 months
  Measure the lateral curvature by Scolioscan. The changes of spinal deformity over a period of 6 months will be evaluated through the sonography.

SECONDARY OUTCOMES:
Contour control | 6 months
  Measure the contour asymmetry by 3D body scanner. The changes of contour asymmetry over a period of 6 months will be evaluated by the 3D scanning images.
Back muscle activity | 6 months
  Measure the back muscle activity signals by the surface electromyography (sEMG) of back muscle. The changes of sEMG of back muscle over a period of 6 months will be evaluated.
Interface pressure of the functional intimate apparel | 2 hours after wearing the functional intimate apparel and 6 months
  Measure the garment interface pressure by the Pliance pressure sensor. The bio-mechanics of the functional intimate apparel are assessed by the changes of pressure distribution.
Health-related quality of life (EQ-5D-5L) | 6 months
  Measure the quality of life by the validated questionnaire, Euroqol (EQ-5D-5L) .The descriptive system comprises 5 dimensions in 5 questions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 0-no problems, 1-slight problems, 2-moderate problems, 3-severe problems and 4-extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number by summed that describes the patient's health state.Total score are ranged from 0 to 20. The higher values represent a worse outcome.
Health-related quality of life (SRS-22) | 6 months
  Measure the quality of life by the validated questionnaire, SRS-22. The questionnaire consists of 22 questions and each question has 5 levels. The SRS-22r measures quality of life across 5 domains - Function (5 questions), Pain (5 questions) Self-Image (5 questions), Mental Health (5 questions), Satisfaction/Dissatisfaction (2 questions). The maximum score in each domain is 5 and minimum score is 1, with higher scores representing greater patient quality of life. The scores of each questions are summed to compute a total score. Total score are ranged from 22 to 110.The higher values represent a better outcome.
Patients' perception of self-image (TAPS) | 6 months
  Measure the subjective impression of trunk deformity by the calidated questionnaire, Trunk Appearance Perception Scale (TAPS). The TAPS includes 3 sets of figures that depict the trunk from 3 viewpoints: looking toward the back, looking toward the head with the patient bending over and looking toward the front. Drawings are scored from 1 (greatest deformity) to 5 (smallest deformity), and a mean score is obtained. The mean score are ranged from 1 to 5. The higher mean scores represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Yip, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China